CLINICAL TRIAL: NCT04156685
Title: An Open-label, Rendomized, Single-dose Crossover Study to Evaluate the Pharmacokinetics, Safety and Tolerability of CKD-387 in Healthy Subjects.
Brief Title: Pharmacokinetics, Safety and Tolerability of CKD-387 10/500mg BE Phase1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A84_07BE1908
Record Dates: First submitted 2019-11-06; First posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Type2 Diabetes Mellitus
Keywords: Type2 Diabetes Mellitus; CKD-387

STUDY DESIGN:
Intervention Model Description: 2 part, 2x2 crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PartA, Treatment-1 (Experimental): Period 1 : Reference drug Period 2 : Test drug
  Interventions: Drug: Part A, Reference (D635 10/500mg, Astrazeneca)
- PartA, Treatment-2 (Experimental): Period 1 : Test drug Period 2 : Reference drug
  Interventions: Drug: Part A, Reference (D635 10/500mg, Astrazeneca)
- PartB, Treatment-1 (Experimental): Period 1 : Reference drug Period 2 : Test drug
  Interventions: Drug: Part B, Reference (D635 10/500mg, Astrazeneca)
- PartB, Treatment-2 (Experimental): Period 1 : Test drug Period 2 : Reference drug
  Interventions: Drug: Part B, Reference (D635 10/500mg, Astrazeneca)

INTERVENTIONS:
Drug: Part A, Reference (D635 10/500mg, Astrazeneca) — Once a day. Under fasting condition
  Other Names: PartA, Test(CKD-387 10/500mg)
  Arms: PartA, Treatment-1
Drug: Part A, Reference (D635 10/500mg, Astrazeneca) — Once a day. Under fasting condition
  Other Names: PartA, Test(CKD-387 10/500mg)
  Arms: PartA, Treatment-2
Drug: Part B, Reference (D635 10/500mg, Astrazeneca) — Once a day. Under fed condition
  Other Names: PartB, Test(CKD-387 10/500mg)
  Arms: PartB, Treatment-1
Drug: Part B, Reference (D635 10/500mg, Astrazeneca) — Once a day. Under fed condition
  Other Names: PartB, Test(CKD-387 10/500mg)
  Arms: PartB, Treatment-2

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, safety and tolerability of CKD-387

DETAILED DESCRIPTION:
An open-label, randomized, single-dose crossover study to evaluate the pharmacokinetics, safety and tolerability of CKD-387 in helalthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult older than 19 years and less than 45 years at the time of screening.
2. BMI 18.5~29.9 kg/m2 and body weight more than 50kg.
3. Subjects who have consented to the use of appropriate double- pregnancy contraceptive methods up to one months after the last investigational product and not to provide sperm for men.
4. Subjects who sign on an informed consent form willingly.

Exclusion Criteria:

1. Subjects who have a clinically significant disease or medical history such as respiratory, hepatic, kidneys, blood, gastrointestinal, endocrine, immune system, skin, nervous and mental disease.
2. Subjects who have acute disease within 28 days prior to the first administration.
3. Subjects who have history that may affect the ADME.
4. Subjects who have medical history or medical abuse history of hypersensitivity from SGLT inhibitors or Biguanides including Metformin or other medications(Aspirin, Antibiotics etc.).
5. Subjects who have clinically significant chronic disease.
6. Subjects with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose mal-absorption.
7. Subjects whose laboratory test result are same as below;

   * AST,ALT > UNL(Upper Normal Limit)x3
   * Fasting glucose level out of 70-125mg/dl
   * Creatinine clearance is lower than 80mL/min which is calcuated by Cockcroft-Gault formulation.
   * QT>450msec
   * Positive urine hCG(female).
8. Subjects whoes blood pressure exceeds out of normal range as below at screening.

   * SBP : over 100mmHg, under 160mmHg
   * DBP : over 60mmHg, under 100mmHg
9. Subjects who have been found to be positive in serological tests(HBs antigen, HCV antibody and HIV antibody).
10. Subjects who took ETC(Ethical Drug), oriental medicine within 2 weeks prior to the first administration of investigational products.
11. Subjects who took OTC(Over-the-counter Drug, including korean galenical drug) within 10 days prior to the first administration of investigational products.
12. Subjects who have allergic disease which has clinical significance(But, light allergic rhinitis and ligth allergic dermatitis which do not need medication is exceptional).
13. Subjects who can not eat standard meals provided by the institution.
14. Subjects who donated whole blood within 60 days, donated the blood components within 20 days prior to the first administration of investigational products.
15. Subjects who received blood transfusion within 30 days prior to the first administration of investigational products.
16. Subjects who were participated in the other clinical trial within 90 days prior to the first administration of investigational products.
17. Subjects who took medication for the induction and inhibition of metabolizing enzymes such as barbiturate drugs within 6months prior to the first administration of investigational products.
18. Subjects who have had abnormal diets that can affect the ADME of the drug within 30 days prior to the first administration of investigational products. (Ingestion of grapefruit juice>1L/day or Caffein>5Cups/day).
19. Subjects who have took regular alcohol(alcohol>30g/day) prior to the first administration of investigational products.
20. Subjects who smoked more than 10 cigarettes per day prior 3months to the first administration of investigational products or cannot discontinue smoking during the clinical trial.
21. Subjects who is determined unsuitable to participate in this clinical trial by the investigator.
22. Lactating Women.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Part A : Cmax under fasting condition | 0(predose)~48 hours
  Maximum concentration of the dapagliflozin
Part A : Cmax under fasting condition | 0(predose)~48 hours
  Maximum concentration of the metformin
Part A : AUClast under fasting condition | 0(predose)~48 hours
  Area Under Curve(last) of the dapagliflozin
Part A : AUClast under fasting condition | 0(predose)~48 hours
  Area Under Curve(last) of the metformin
Part B : Cmax under fed condition | 0(predose)~48 hours
  Maximum concentration of the metformin
Part B : AUClast under fed condition | 0(predose)~48 hours
  Area Under Curve(last) of the metformin

SECONDARY OUTCOMES:
Part A : AUCinf under fasting condition | 0(predose)~48 hours
  Area Under Curve(infinit) of the dapagliflozin
Part A : AUCinf under fasting condition | 0(predose)~48 hours
  Area Under Curve(infinit) of the metformin
Part A : Tmax under fasting condition | 0(predose)~48 hours
  Time of maximum concentration of the dapagliflozin
Part A : Tmax under fasting condition | 0(predose)~48 hours
  Time of maximum concentration of the metformin
Part A : t1/2 under fasting condition | 0(predose)~48 hours
  Half life of the dapagliflozin
Part A : t1/2 under fasting condition | 0(predose)~48 hours
  Half life of the metformin
Part B : AUCinf under fed condition | 0(predose)~48 hours
  Area Under Curve(infinit) of the metformin
Part B : Tmax under fed condition | 0(predose)~48 hours
  Time of Maximum concentration of the metformin
Part B : t1/2 under fed condition | 0(predose)~48 hours
  Half life of the metformin

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Young Park, M.D, Ph.D, Principal Investigator — Korea University Anam Hospital / Seoul, Seongbuk-Gu, South Korea
Locations (1):
- Korea University Anam Hospital, Seoul, Seongbuk-Gu, South Korea